CLINICAL TRIAL: NCT03749564
Title: Examining the Influence of Opioid Use on the Effects of Spinal Manipulative Therapy for Low Back Pain: Administrative Supplement to UH3AT009293 - Optimization of Spinal Manipulative Therapy (SMT) Protocols
Brief Title: Influence of Opioid Use on the Effects of Spinal Manipulative Therapy for Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 restrictions on research activities
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Julie Fritz, Professor, University of Utah
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 59006084
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Low Back Pain; Opioid Use
Keywords: Spinal Manipulative Therapy; Optimization
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Factorial design examining the outcomes of SMT with varying combinations of co-interventions.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Design precludes blinding of patients or care providers. Research personnel conducting outcomes assessments and the principal investigator are blind to participants' group assignment throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SMT Only (Experimental): All patients receive 2 SMT sessions in the first week.
  Interventions: Behavioral: SMT
- SMT extended (Experimental): All patients receive 2 SMT sessions in the first week. This arm also involves 6 additional SMT sessions. Each SMT session is conducted as described previously.
  Interventions: Behavioral: SMT; Behavioral: Extended SMT
- SMT with Activation Exercises (Experimental): All patients receive 2 SMT sessions in the first week.
  This arm receives 6 additional sessions of activation exercises.
  Interventions: Behavioral: SMT; Behavioral: Activation Exercises
- SMT with Mobilizing Exercises (Experimental): All patients receive 2 SMT sessions in the first week.
  This arm involves 6 additional sessions of mobilizing exercise.
  Interventions: Behavioral: SMT; Behavioral: Mobilizing Exercises
- SMT with Mobilizing and Activation Exercises (Experimental): All patients receive 2 SMT sessions in the first week.
  This arm involves 6 additions sessions including both activation and mobilizing exercises.
  Interventions: Behavioral: SMT; Behavioral: Activation Exercises; Behavioral: Mobilizing Exercises
- SMT extended with Mobilizing Exercises (Experimental): All patients receive 2 SMT sessions in the first week.
  This arm includes 6 additional sessions including both SMT and mobilizing exercises.
  Interventions: Behavioral: SMT; Behavioral: Mobilizing Exercises; Behavioral: Extended SMT
- SMT extended with Activation Exercises (Experimental): All patients receive 2 SMT sessions in the first week.
  This arm includes 6 additional sessions including both SMT and activation exercises.
  Interventions: Behavioral: SMT; Behavioral: Activation Exercises; Behavioral: Extended SMT
- SMT extended with Mobilizing and Activation Exercises (Experimental): All patients receive 2 SMT sessions in the first week.
  This arm includes 6 additional sessions including SMT, activation and mobilizing exercises.
  Interventions: Behavioral: SMT; Behavioral: Activation Exercises; Behavioral: Mobilizing Exercises; Behavioral: Extended SMT

INTERVENTIONS:
Behavioral: SMT — The subject is supine. The clinician stands opposite the side to be manipulated and side-bends the subject away from the side to manipulate. The side to be manipulated is the more painful. If the subject cannot identify a more painful side the clinician selects a side. The clinician rotates the subject, and delivers a high-velocity, low-amplitude (HVLA) thrust to the pelvis in a posterior/inferior direction. The clinician notes if a cavitation (ie, a "pop") occurred. If it does, SMT treatment is complete. If no cavitation occurs, the subject is repositioned and SMT is performed again. If no cavitation occurs on the second attempt, the clinician manipulates the opposite side. A maximum of 2 attempts per side is permitted. If no cavitation is noted by that time, SMT treatment is complete. Substitution with a side-posture HVLA technique is allowed if the preferred technique is not possible due to subject preference or comfort.
  Other Names: spinal manipulative therapy
Behavioral: Activation Exercises — Activation exercises are designed to facilitate use of the lumbar multifidus muscle. Exercises will begin with isometric multifidus contractions in different positions with clinician feedback and exercises to isometrically co-contract the multifidus and deep abdominal muscles. Subjects will also perform lumbar extensor strengthening exercises shown to produce 20%-50% of multifidus maximum voluntary contraction. Subjects will continue to perform isometric exercises throughout treatment. Subjects will perform their prescribed exercises at treatment sessions and will be instructed to perform the exercises daily on other days.
  Arms: SMT extended with Activation Exercises; SMT extended with Mobilizing and Activation Exercises; SMT with Activation Exercises; SMT with Mobilizing and Activation Exercises
Behavioral: Mobilizing Exercises — Mobilizing exercises include a program of repeated movements progressing into end-ranges of spinal flexion and/or extension shown in past studies to improve ROM and reduce spinal stiffness. Patients will be instructed in mid-range exercises and will be further assessed for a directional preference. A directional preference is present if movement in a particular direction decreases LBP intensity or causes symptoms to centralize towards the midline. If a subject has a directional preference he or she will be prescribed exercises specifically in that direction along with mid-range exercise. Otherwise the subject will be assigned exercises moving into either flexion or extension based on the clinician's discretion. Subjects will perform their prescribed exercises at treatment sessions and will be instructed to perform the exercises daily on other days.
  Arms: SMT extended with Mobilizing Exercises; SMT extended with Mobilizing and Activation Exercises; SMT with Mobilizing Exercises; SMT with Mobilizing and Activation Exercises
Behavioral: Extended SMT — Additional 6 SMT sessions provided
  Arms: SMT extended; SMT extended with Activation Exercises; SMT extended with Mobilizing Exercises; SMT extended with Mobilizing and Activation Exercises

SUMMARY:
This project is a supplement to the parent project (UH3AT009293) entitled "Optimization of Spinal Manipulative Therapy (SMT) Protocols". The goal of the parent project is to examine strategies to optimize SMT treatment protocols for patients with low back pain (LBP). The parent project is investigating mechanistic and clinical outcomes of SMT combined with varying co-interventions. This supplemental project will examine the impact of opioid use on these outcomes.

DETAILED DESCRIPTION:
This supplement expands the parent research project to include three additional Aims and the recruitment of the 70 additional participants. The additional participants will undergo the same assessment and intervention procedures outlined in the parent project to permit leveraging the full cohort to evaluate the supplemental Aims.

The overall objective is to examine the impact of opioid use on patient-centered and mechanistic outcomes related to SMT and explore the impact on SMT followed by various co-interventions. The goal of this research is to better tailor SMT protocols to optimize outcomes for patients with LBP who are opioid users and facilitate efforts to reduce reliance on opioid pain management among those with LBP. Accomplishing this goal will facilitate future research evaluating the efficacy of non-pharmacologic alternative pain management strategies for individuals with LBP.

Specific Aims to be addressed through this supplement are:

1. Compare baseline psychological, mechanistic and LBP-related characteristics between sub-groups of participants with LBP based on opioid use.
2. Examine the association of opioid use with changes in mechanistic and patient-centered outcomes between a baseline assessment and subsequent assessment after 1-week and completion of a 2-session SMT intervention protocol.
3. Explore the moderating effects of opioid use on mechanistic and patient-centered outcomes obtained 4 weeks following SMT intervention with varied co-intervention components.

Examining these aims as a supplement to the parent project will allow evaluation of whether or not opioid use impacts short-term mechanistic and patient-centered outcomes of SMT (Aim 2), and will explore if the longer-term effects of the three co-interventions differ between opioid users and non-users. (Aim 3). This research will also compare baseline characteristics between participants who are or are not opioid users (Aim 1).

ELIGIBILITY:
Inclusion Criteria:

* Pain between the 12th rib and buttocks with or without symptoms into one or both legs, which, in the opinion of the examiner, originate from the lumbar region.
* Age 18 - 60 years
* Oswestry disability score > 20%
* Self-reported

Exclusion Criteria:

* Prior surgery to the lumbosacral spine
* Currently pregnant
* Currently receiving mind-body or exercise treatment for LBP from a healthcare provider (e.g., chiropractic, physical therapy, massage therapy, etc.)
* Neurogenic signs including any of the following: positive ipsi- or contra-lateral straight leg raise test; reflex, sensory, or strength deficit in a pattern consistent with lumbar nerve root compression

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Oswestry | 1 week
  The Oswestry Index measures back pain-related disability. The scale contains 10 items with a final score ranging from 0-100. Higher numbers indicate more disability.
Pain intensity: 0-10 numeric pain rating | 1 week
  A 0-10 numeric pain rating is used to assess pain intensity. Higher numbers indicate greater pain intensity.

SECONDARY OUTCOMES:
Multifidus Activation | Baseline, 1-week, 4-weeks, 3 months
  Multifidus activation wis measured with brightness-mode ultrasound images using a 60mm, 2-5 MHz curvilinear array. The subject is prone. The ultrasound transducer is placed just lateral to midline and angled medially until a parasagittal view of the multifidus is obtained. Images are acquired at each level with the multifidus at rest and during submaximal contraction elicited by the subject lifting the contralateral arm about 2 inches while holding a weight proportional to body weight. Three images in each state are acquired and averaged. Offline multifidus thickness measures are obtained from the distance between the posterior-most aspect of the facet joint inferiorly and the plane between the multifidus and thoracolumbar fascia superior. Muscle activation is calculated as the change in thickness at rest and submaximal contraction and expressed in mm.
Spinal Stiffness | Baseline, 1-week, 4-weeks, 3 months
  Spinal stiffness is assessed with a mechanically-assisted indentation device over the spinous processes. Indentation involves advancement of the probe from a 5 N pre-load to 60 N final load maintained for 1 second, then the probe raises automatically. Three indentation trials are performed with mean values used for analysis. Indentation data (force and displacement) are used to calculate stiffness variables. Global stiffness (N) is calculated as the slope of the force displacement curve between 5 - 60 N, representing stiffness of underlying tissues during indentation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Department of Physical Therapy, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No